CLINICAL TRIAL: NCT04553614
Title: Home-based High Intensity Interval Training is Effective in a Primary Care Setting for at Risk Individuals: A Multidisciplinary Approach Evaluating Health and Perceived Barriers to Exercise
Brief Title: Home-based HIIT in a Primary-care Setting for at Risk Individuals: A Multidisciplinary Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Collaborators: Loughborough University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Home-HIIT and ERS
Record Dates: First submitted 2020-09-04; First posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Risk Factor, Cardiovascular
Keywords: HIIT; Cardiorespiratory fitness; Heart Rate; Feasibility; Exercise; Exercise Prescription; Primary Health Care; Humans
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Referral Scheme (Active Comparator): The active Sefton (AS_ERS) is a traditional exercise referral programme providing highly discounted access to council operated leisure centres and a number of partner gyms. Within this access patients will have access to gym and swimming facilities (£2 per visit) and exercises classes (£3 per visit). During the patients first meeting with their LDO a progressive personalised exercise programme will be developed. Following this the patient will attend their local gym or leisure centre for an induction with a staff member(£7 one off fee), enabling them to attend the centre at any time and complete the designed exercise programme. All exercise programmes will be different, but in general will include moderate intensity exercise on gym equipment (treadmill, ergometer etc.) and some basic resistance training. Patients may replace these gym sessions with exercises classes run by the facility. Patients will be encouraged to exercise 3-5 time per week.
  Interventions: Other: Control
- Home-based HIIT (Experimental): Participants will be instructed to complete each training session in a place of their choosing. The programme involves repeated 1 minute bouts of simple on the spot movements interspersed with 1 minute of rest. During the intervals participants will be advised to reach a heart rate of approx. 90% of their predicted maximum heart rate (220-age). The 1 minute interval will be split between 2 consecutive 30 second exercises. The research team have a library of 18 exercises, with 9 suggested exercise pairs. The participant will be advised to complete 4 intervals during weeks 1 and 2, with the number of intervals increasing by 1 every 2 weeks (maximum of 9 intervals). The participant will be advised to train 3x per week.
  Interventions: Behavioral: Home-based HIIT

INTERVENTIONS:
Behavioral: Home-based HIIT — Home-based HIIT uses body-weight equipment free exercises. Participants complete all exercise in their own own at a time of their choosing. This potentially removes many of the barriers preventing at risk-individuals from engaging with the current exercise referral scheme, such as cost, time or intimidating gym environment.
  Arms: Home-based HIIT
Other: Control — Usual exercise referral scheme procedure.
  Arms: Exercise Referral Scheme

SUMMARY:
The prevalence of chronic inactivity related diseases including obesity, insulin resistance and type 2 diabetes mellitus has reached global epidemic proportions. Exercise training is a clinically proven primary intervention that delays and in many cases prevents health burdens. Therefore, many health authorities and local councils run exercise referral schemes for individuals with elevated disease disk. However, a number of barriers to successful completion of traditional exercise referral schemes exist.

This study aims to investigate the use of a home-based high intensity interval training programme as a potential exercise referral scheme activity to overcome many of the barriers to successful exercise referral scheme adherence and uptake.

200 people referred to the Active Sefton (Sefton Council) exercise referral scheme will be recruited and randomised to one of the two exercise groups (existing Active Sefton Scheme gym based training or home-based HIT). All participants will have access to the normal Active Sefton support mechanisms, but the training programme followed will be different. Before and after 12 weeks of training volunteers will participate in testing to assess changes in aerobic fitness, physical activity, vascular function, insulin sensitivity, body composition and psychological well-being. A 3 month follow up will also be completed to investigate the long term consequences on these variables.

DETAILED DESCRIPTION:
Randomisation - During the pre-intervention testing session participants will be randomised to either the home-based HIT group (HB_HIT)(n=100) or Active Sefton Exercise Referral Scheme (AS_ERS)(n=100). To control for the potential confounding effects of gender and location, stratified randomisation will be completed. Randomisation will be completed with a random number generator. Participant randomisation will take place during Pre-Intervention Testing.

Recruitment - Participants will be recruited via the AS_ERS. Following referral to the Active Sefton Scheme by their GP, all patients will be sent an invitation letter by the Active Sefton team. The research team will add a short letter outlining the study to patients. All Patients who chose to participate in the Active Sefton Scheme will meet with an Active Lifestyle Development Officer (LDO). During this session the LDO will discuss the study with patients. Interested patients will be given a participant information sheet, and their contact details (email and/or phone) will be given to the Liverpool John Moores University (LJMU) research team. These details will be used to contact the patient to discuss the study further. Should the patient still want to participate a Pre-Intervention Testing session will be organised.

If patients consent to the study the research team will inform Active Sefton with information on the exercise programme the participant has been randomised too.

Protocol and plan of investigation

Pre-Intervention Testing - Participants will attend an experimental trial commencing between 6am and 10am, lasting ̴ 3.15h. Participants will be fasted overnight and instructed to abstain from caffeine, alcohol and moderate/ vigorous exercise the day before testing.

During this meeting participants will have the opportunity to ask any questions about the study. Participants will then be asked to give written consent (participants may wish to take longer to decide and this testing session will be rearranged if necessary). If consent is given participants will complete a number of health measurements.

Firstly, following 20 minutes supine rest central artery stiffness will be measured using a Sphygmocor system. A blood pressure recording will be taken at the brachial artery and an ECG waveform obtained. A tonometer will then be applied with gentle pressure at the femoral and carotid arteries (thigh/neck) to measure aortic pulse wave velocity (a measure of arterial stiffness).

Insulin sensitivity will be measured through an OGTT. A cannula will be placed into a forearm vein of one arm and will be used to obtain repeated blood samples. A resting blood sample (25ml) will be taken immediately before consumption of a 25% glucose beverage (75g of glucose). Following this further blood samples (5ml) will be collected 15, 30, 45, 60, 90 and 120 minutes after glucose ingestion. During the OGTT participants will complete a number of other measures.

Firstly, participants will complete a questionnaire pack to assess psychological well-being and self- report physical activity. The pack will include the International Physical Activity Questionnaire (IPAQ), General positive and negative affect (PANAS), Subjective Vitality Scale (SVS), Health Perception (item from Medical Outcomes survey: MOS SF-36), Satisfaction with Life Scale (SWLS), Behavioural Regulations to Exercise (BREQ-3), Adapted Perceived Competence (PCS). Anthropometric measures will be taken (height, weight, waist-to-hip ratio). Body composition will then be measured using dual-energy X-ray absorptiometry scanning.

Finally, once the OGTT is completed an incremental maximal aerobic capacity test (VO2max) to volitional exhaustion will be conducted on a cycle ergometer. Throughout the test, measures of oxygen uptake, blood pressure and heart rate will be taken. This test will allow us to determine maximal oxygen uptake (VO2max) and maximal power output (Wmax). Following the test heart rate recovery kinetics will be monitored.

Post-Intervention Testing 3-7 days after their last training session participants will attend the laboratory for a post-intervention testing session. This session will be identical in all respects to the pre-intervention testing session.

Version 1 15/12/16

3-Month Follow-up - 3-months after post-intervention testing participants will attend a final testing session identical in all respects to the pre-intervention testing session.

Home-based HIT - Participants will be provided with a training guide containing information on the exercises and a suggested programme. The programme will also be explained during the Pre-Intervention Testing session. Participants will be instructed to complete each training session in a place of their choosing. The programme involves repeated 1 minute bouts of simple on the spot movements interspersed with 1 minute of rest. During the intervals participants will be advised to reach a heart rate of approx. 90% of their predicted maximum heart rate (220-age). The 1 minute interval will be split between 2 consecutive 30 second exercises. The research team have a library of 18 exercises, with 9 suggested exercise pairs. The participant will be advised to complete 4 intervals during weeks 1 and 2, with the number of intervals increasing by 1 every 2 weeks (maximum of 9 intervals). The participant will be advised to train 3x per week.

Active Sefton Exercise Referral Scheme - The AS_ERS is a traditional exercise referral programme providing highly discounted access to council operated leisure centres and a number of partner gyms. Within this access patients will have access to gym and swimming facilities (£2 per visit) and exercises classes (£3 per visit). During the patients first meeting with their LDO a progressive personalised exercise programme will be developed. Following this the patient will attend their local gym or leisure centre for an induction with a staff member(£7 one off fee), enabling them to attend the centre at any time and complete the designed exercise programme. All exercise programmes will be different, but in general will include moderate intensity exercise on gym equipment (treadmill, ergometer etc.) and some basic resistance training. Patients may replace these gym sessions with exercises classes run by the facility. Patients will be encouraged to exercise 3-5 time per week. Participants will be given a training diary by the study team where they will be encouraged to write details of the training sessions completed.

3-Month Follow-up- Following the 12 week study intervention participants will be given the opportunity to complete the alternative intervention (HB_HIT or AS_ERS). Participants wanting to complete the HB_HIT programme will be given a training guide and have the intervention explained to them by the research team. Participants wanting to complete the AS_ERS will be given discounted access to their local leisure centre for 12 weeks (see above) and a gym induction will be arranged for them by their LRO. Neither group will have contact with the Active Sefton Team, including LDO, during this 3-month period.

Heart Rate Monitoring - All Participants (HB_HIT and AS_ERS) will be given a polar H7 Bluetooth heart rate monitor. Participants will be advised to wear this monitor during all training sessions. The monitor will provide a measure of training intensity for the AS_ERS group, and compliance with the suggested heart rate target in the HB_HIT group.

Participants will be asked to download Polar Beat to their smartphone (a free Android and IOS app). This app will be used to monitor heart rate during the training sessions. In addition, participants will be given a login email address and password for Polar Flow (www.polar.flow.com), a cloud storage site run by Polar for the storage and analysis of heart rate data. All heart rate data measured during training sessions will be uploaded to Polar Flow. This will allow the research team to investigate training intensity achieved during all sessions.

Active Sefton Support - Throughout the study all participants (AS_ERS and HB_HIT) will receive the normal support provided by the Active Sefton Scheme. This takes the form of 3 sessions with an LDO. These sessions will be pre, mid (6 weeks) and following the exercise interventions. The LDO will be informed of the exercise programme conducted by the participant, enabling them to provide program specific support to patients.

ELIGIBILITY:
Inclusion Criteria:

Referred to Active Sefton Exercise Referral scheme by a GP Aged 18-65

Referral criteria:

High blood pressure Angina (treated and stable) Mental Health issues (anxiety/ stress/ depression) Previous Heart attack or heart surgery (not under current investigation) Diabetes type 1 or 2 Impaired glucose tolerance Overweight/ obese (BMI >30)

Exclusion Criteria:

* Aged <18 or >65
* Cardiac rehab patient
* In order to take part participants should have a good grasp of spoken English
* Blood pressure >180/100 and/or uncontrolled or poorly controlled hypertension
* Currently prescribed Beta-blockers
* Cardiomyopathy
* Uncontrolled tachycardia
* Cardiac arrhythmia
* Valvular heart disease
* Aneurysms
* Diabetes and 1 of the following:

  * Aged >35
  * Type 2 diabetes mellitus >10 yr duration
  * Type 1 diabetes mellitus >15 yr duration
  * Hypercholesterolemia (total cholesterol >6.2 mmol/l)
  * Hypertension (systolic blood pressure >140 or diastolic >90 mm Hg)
  * Smoking
  * Family history of coronary artery disease (CAD) in first-degree relative <60 yr o Presence of microvascular disease
  * Peripheral vascular disease
  * Autonomic neuropathy
* Uncontrolled (drug resistant) epilepsy - failed to become (and stay) seizure free following trials of two seizure medications.
* History of falls or dizzy spells in the last 12 months
* Excessive or unexplained breathlessness on exertion
* Uncontrolled or poorly controlled asthma (severe COPD) - Limitation in performing day-to-day activities, weekly nocturnal symptoms and awakening, more need for rescue medications, lung function (FEV1) < 80%, three or more asthma attacks per year
* Pregnant or breast feeding or becomes pregnant during the study
* End stage renal disease
* Awaiting medical investigation
* Severe mental health condition
* Any other medical condition or condition that would make them unsuitable for an exercise programme.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory fitness | 3 months
  Incremental exercise test to exhaustion to assess VO2peak

SECONDARY OUTCOMES:
Body composition | 3 months
  via DXA
Insulin Sensitivity | 3 months
  Oral Glucose Tolerance Test
Exercise Adherence | 3 months
  Participants to record all complete exercise sessions using a Bluetooth compatible heart rate monitor, linked to cloud data storage. Research team will have access to cloud storage to assess the number of exercise sessions completed.

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool John Moores University, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hesketh K, Jones H, Kinnafick F, Shepherd SO, Wagenmakers AJM, Strauss JA, Cocks M. Home-Based HIIT and Traditional MICT Prescriptions Improve Cardiorespiratory Fitness to a Similar Extent Within an Exercise Referral Scheme for At-Risk Individuals. Front Physiol. 2021 Nov 10;12:750283. doi: 10.3389/fphys.2021.750283. eCollection 2021. PMID 34858205